CLINICAL TRIAL: NCT03805620
Title: Synergistic Effects of Combined Physical-cognitive Training on Cognitive Function in Individuals With Mild Cognitive Impairment (MCI): A Randomized Controlled Trial
Brief Title: Effects of Combined Physical-cognitive Training on Cognitive Function in MCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Somporn Sungkarat, Associate Professor, Chiang Mai University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: AMS-CMU
Record Dates: First submitted 2019-01-07; First posted 2019-01-15 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Mild Cognitive Impairment
Keywords: mild cognitive impairment; combined physical-cognitive training; BDNF; mitochondrial function; cognitive function
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Physical Conditioning, Human; Cognitive Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Phys Group (Active Comparator): physical training group
  Interventions: Other: Physical training
- Cog Group (Active Comparator): cognitive training group
  Interventions: Other: Cognitive training
- Phys-Cog Group (Experimental): combined physical-cognitive training group
  Interventions: Other: Combined physical-cognitive training
- Con Group (No Intervention): educational control group

INTERVENTIONS:
Other: Combined physical-cognitive training — combined physical-cognitive training
  Arms: Phys-Cog Group
Other: Physical training — Multi-component physical exercise
  Arms: Phys Group
Other: Cognitive training — cognitive training
  Arms: Cog Group

SUMMARY:
The present study aims to investigate the effects of combined physical-cognitive training on cognitive function as well as peripheral BDNF level and mitochondrial function of individuals with MCI. It is hypothesized that: 1) the combined physical-cognitive training program will be superior to the physical and cognitive training program alone; and 2) the degree of cognitive improvement will be positively correlated with the improvement of plasma BDNF and mitochondrial function.

DETAILED DESCRIPTION:
Recent research suggests that the benefits of combined physical-cognitive training may be greater than either physical or cognitive training alone. Nevertheless, this synergistic effect has been demonstrated mainly in cognitively intact older adults. Studies examining the effects of combined physical-cognitive training in older adults with MCI are scarce and show mixed results. Moreover, few studies have determined the effects of the combined training on peripheral brain-derived neurotrophic factor (BDNF) and mitochondrial function. Thus, the present study aims to investigate the effects of combined physical-cognitive training on cognitive function as well as peripheral BDNF level and mitochondrial function of individuals with MCI. The present study will provide insight into the interplay among the training program, peripheral BDNF concentration, mitochondrial function, and cognitive function. Importantly, the findings will have clinical implication regarding the training program that is feasible and effective in improving cognitive function of older adults with MCI which ultimately will have great impact on public health as this population is at high risk of progression to AD.

ELIGIBILITY:
Inclusion Criteria:

* meet criteria for mNCD (mild neurocognitive disorders), previously known as MCI, based on the recent DSM-V (Diagnostic Statistical Manual-V) criteria
* comprehend instructions and willing to participate
* able to comply with the study schedule and procedures
* not taking any medications for their cognition and not planning to start medications during the study trial

Exclusion Criteria:

* presence of medical conditions that would be unsafe to exercise
* diagnosed with other neurological conditions (e.g. Parkinson's disease, Stroke, Multiple Sclerosis, AD) that affect cognition and mobility
* presence of depressive symptoms
* presence of acute or/and chronic disease that could not be controlled (e.g. Arthritis, Asthma, Hypertension, Diabetes mellitus, Coronary artery disease)
* exercise regularly (at least 30 min/day, 3 days/week)

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-06-28 (Actual)

PRIMARY OUTCOMES:
change from baseline Alzheimer's Disease Assessment- cognitive subscale at 3 months | 3 months
  Alzheimer's Disease Assessment-cognitive subscale will be assessed at baseline and 3 months. The total scores range from 0-70, with higher scores (≥ 18) indicating greater cognitive impairment.
change from baseline Rey auditory verbal learning score at 3 months | 3 months
  Memory will be assessed using Rey auditory verbal learning test.
change from baseline Trail Making B-A score at 3 months | 3 months
  Executive function will be assessed using Trail Making Test part B-A.
change from baseline brain-derived neurotrophic factor level at 3 months | 3 months
  Level of plasma brain-derived neurotrophic factor (BDNF) will be determined.

SECONDARY OUTCOMES:
change from baseline Digit Span score at 3 months | 3 months
  Attention will be assessed using Digit Span forward-backward test.
change from baseline stepping response time at 3 months | 3 months
  Processing speed will be measured using stepping response time.
change from baseline time to complete Timed Up and Go at 3 months | 3 months
  Functional ability will be assessed using time to complete Timed Up and Go (TUG).
change from baseline physiological profile assessment score at 3 months | 3 months
  Fall risk will be assessed using the physiological profile assessment. The test consists of five sensorimotor and balance measures including visual contrast sensitivity, proprioception, quadriceps muscle strength, hand reaction time, and postural sway. The five PPA components are weighted to compute a composite z-score distribution with high scores indicating increased fall risk.
change from baseline cellular oxidative stress level at 3 months | 3 months
  Mitochondrial function will be determined from cellular oxidative stress level

CONTACTS AND LOCATIONS:
Overall Officials: Somporn Sungkarat, PhD, Principal Investigator — Chiang Mai University
Locations (1):
- Faculty of Associated Medical Sciences, Chiang Mai University, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: No